CLINICAL TRIAL: NCT01790984
Title: How Does Dietary Carbohydrate Influence the Formation of an Atherogenic Lipoprotein Phenotype?
Brief Title: How Does Dietary Carbohydrate Influence the Formation of an Atherogenic Lipoprotein Phenotype (ALP)?
Acronym: CHOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruce A. Griffin (Other)
Collaborators: Imperial College London (Other); University of Cambridge (Other)
Responsible Party: Sponsor-Investigator, Bruce A. Griffin, Professor of Nutritional Metabolism, University of Surrey
Organization: University of Surrey (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RN0172 A/B; BB/G009899/1 (Other Grant/Funding Number: BBSRC)
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Results first posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: Sugars, Fatty liver, Lipoprotein kinetics, Triglycerides
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High sugar low starch diet (Experimental): A high sugar, low starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with low sugar to starch content, with foods containing a high sugar to starch content to reach a target ratio of starch to sugar of 1:1.2
  Interventions: Other: High sugar low starch diet; Other: Low sugar high starch diet
- Low sugar high starch diet (Experimental): A high sugar, low starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with a high sugar to starch content, with foods containing a low sugar to starch content to reach a target ratio of starch to sugar of 5:1
  Interventions: Other: High sugar low starch diet; Other: Low sugar high starch diet

INTERVENTIONS:
Other: High sugar low starch diet
Other: Low sugar high starch diet

SUMMARY:
The hypothesis of this study is that a diet high in sugars will increase abnormalities in blood lipids which are associated with increased cardiovascular disease risk, relative to a diet which is low in sugar. We predict that this potentially adverse effect of dietary sugars on blood lipids will be more pronounced in people with a raised level of stored fat inside their liver, as compared to people with a low level of stored fat.

DETAILED DESCRIPTION:
This study aims to determine the metabolic mechanism(s) by which dietary extrinsic sugars (sucrose and fructose), promote the formation of a high risk dyslipidaemia, known as an atherogenic lipoprotein phenotype (raised plasma triglyceride, low HDL and predominance of small, dense LDL), in men with raised cardio-metabolic risk and percentage of liver fat, as determined by magnetic resonance spectroscopy (MRS). The study examined the impact of diets high and low in extrinsic sugars, on the metabolism of lipids and lipoproteins in vivo, of two groups of men with a high (>10%)and low (<2%)percentage of liver fat, by the trace-labelling of these lipid moieties with stable isotopes, and detection by gas chromatography mass spectrometry. The study had a two-way cross-over design, with two, 12 week dietary interventions separated by a six week wash-out period. The dietary intervention with high and low sugars was achieved by a dietary exchange with supermarket foods, which were consumed within the homes of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Male gender,
* Increased cardio-metabolic risk ('RISCK' criteria Jebb et al (2010) Am J Clin Nutr 92, 748-758).
* Apo E3E3 genotype

Exclusion Criteria:

* Any abnormal result in blood screen (renal and liver function, haematology)
* Diabetes
* Smoker
* Excessive alcohol consumption (>27units/week)
* Medication likely to affect lipid metabolism
* >3kg weight loss in preceding 3 months
* Any medical condition (eg. GI tract, allergies) affecting lipid metabolism or ability to comply with dietary interventions
* Involvement in any other study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Griffin, PhD, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited over a period of 24 months (2009-2011) at the 'CEDAR' Centre for Endocrinology and Diabetes Research, Royal Surrey County Hospital, Guildford, Surrey, United Kingdom.
Pre-assignment Details: Men were selected on the basis of expressing increased cardio-metabolic risk and APOE E3E3 genotype. The men were screened for intracellular hepatic fat by magnetic resonance spectroscopy (MRS) and divided into two groups: low liver fat Controls (<5% liver fat) and non-alcoholic fatty liver disease (NAFLD) with percentage liver fat >5%.
Groups:
- High Sugar / NAFLD: Men with NAFLD (>5% liver fat) on a high sugar diet (25% total energy)
  Please note: This was a randomised cross-over study. The men with NAFLD and Controls were randomised to either diet in the 'First Dietary Intervention (12 weeks)' period, and after the 'Wash-out (4 weeks)' period, crossed-over to the alternate diet in the 'Second Dietary Intervention (12 weeks)' period. This is why the number completing the First Intervention is not the same as the number starting the Second Dietary Intervention.
- High Sugar / Controls: Controls (<5% liver fat) on a high sugar (HS) diet.
  Please note: This was a randomised cross-over study. The men with NAFLD and Controls were randomised to either diet in the 'First Dietary Intervention (12 weeks)' period, and after the 'Wash-out (4 weeks)' period, crossed-over to the alternate diet in the 'Second Dietary Intervention (12 weeks)' period. This is why the number completing the First Intervention is not the same as the number starting the Second Dietary Intervention.
- Low Sugar / NAFLD: Men with NAFLD (>5% liver fat) on a low sugar diet.
  Please note: This was a randomised cross-over study. The men with NAFLD and Controls were randomised to either diet in the 'First Dietary Intervention (12 weeks)' period, and after the 'Wash-out (4 weeks)' period, crossed-over to the alternate diet in the 'Second Dietary Intervention (12 weeks)' period. This is why the number completing the First Intervention is not the same as the number starting the Second Dietary Intervention.
- Low Sugar / Controls: Controls with low liver fat (<5%) on a low sugar diet (5% total energy)
  Please note: This was a randomised cross-over study. The men with NAFLD and Controls were randomised to either diet in the 'First Dietary Intervention (12 weeks)' period, and after the 'Wash-out (4 weeks)' period, crossed-over to the alternate diet in the 'Second Dietary Intervention (12 weeks)' period. This is why the number completing the First Intervention is not the same as the number starting the Second Dietary Intervention.
Period: First Dietary Intervention (12 Weeks)
Arm/Group | High Sugar / NAFLD | High Sugar / Controls | Low Sugar / NAFLD | Low Sugar / Controls
Started | 6 | 8 | 6 | 7
Completed | 5 | 7 | 6 | 7
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Period: Wash-out (4 Weeks)
Arm/Group | High Sugar / NAFLD | High Sugar / Controls | Low Sugar / NAFLD | Low Sugar / Controls
Started | 5 | 7 | 6 | 7
Completed | 5 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Second Dietary Intervention (12 Weeks)
Arm/Group | High Sugar / NAFLD | High Sugar / Controls | Low Sugar / NAFLD | Low Sugar / Controls
Started | 5 | 7 | 6 | 7
Completed | 5 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Entry criteria for the two study groups of men included an APO e3/e3 genotype, and either a high percentage of liver fat of greater than 5% (by volume) = NAFLD (if excess alcohol intake excluded) or low percentage of liver fat of less than 5% ('Control' status) at baseline, before being randomised to the two dietary treatments in a two-way cross-over design.
Groups:
- NAFLD (>5% Liver Fat): Men with non-alcoholic fatty liver disease (NAFLD) n=12
- Controls (<5% Liver Fat): Controls (men without NAFLD <5% liver fat) n=15
- Total: Total of all reporting groups
Arm/Group | NAFLD (>5% Liver Fat) | Controls (<5% Liver Fat) | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (4.7) | 54 (7.3) | 57 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 15 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body weight [Mean (Standard Deviation); unit: kilograms] | 89.7 (7.8) | 89.6 (9.1) | 89.7 (8.4)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 28.8 (1.4) | 28.5 (1.5) | 28.6 (1.4)
Serum cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.90 (0.83) | 5.51 (1.00) | 5.70 (1.00)
Serum triacylglycerol [Mean (Standard Deviation); unit: mmol/L] | 2.05 (0.88) | 1.51 (0.87) | 1.70 (0.90)
Serum glucose [Mean (Standard Deviation); unit: mmol/L] | 5.73 (0.45) | 5.46 (0.45) | 5.58 (0.43)
Serum HDL cholesterol [Mean (Standard Deviation); unit: mmol/L] | 1.35 (0.28) | 1.34 (0.30) | 1.34 (0.29)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 134 (19) | 132 (13) | 133 (16)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 85 (13) | 83 (9) | 85 (11)

OUTCOME MEASURES:

1. Primary Outcome: Production Rate of VLDL-1 Triacylglycerol (TAG)
Description: The in vivo production rate of VLDL-1 TAG, trace-labelled with [1,1,2,3,3-H5] glycerol, measured in units of grams/day.
Time Frame: After (post-diet) two 12 week diets (high sugar versus low sugar) in men with NAFLD (n=11) versus Controls (n=14)
Population: Population consisted of two groups: Group 1: men with non-alcoholic fatty liver disease (NAFLD) raised liver fat (>5%) n=11. Group 2: Controls; men with low liver fat (<5%) n=14.
Measure: Mean (Standard Error); unit: grams/day
Groups:
- High Sugar Diet (12 Weeks) in Men With NAFLD: A high sugar (27% total energy), low starch diet was provided by the exchange of 66% of the participants daily intake of carbohydrate. This was achieved by exchanging foods with a low sugar to starch content, with foods containing a high sugar to starch content to reach a target ratio of starch to sugar 1: 1.2.
- Low Sugar Diet (12 Weeks) in Men With NAFLD: A low sugar (9% total energy), high starch diet was provided by the exchange of 66% of the participants daily intake of carbohydrate. This was achieved by replacing foods with a high sugar to starch content, with foods containing a low sugar to starch content to reach a target ratio of starch to sugar of 5:1
- High Sugar Diet (12 Weeks) in Controls: A high sugar (28% total energy), low starch diet was provided by the exchange of 66% of the participants daily intake of carbohydrate. This was achieved by exchanging foods with a low sugar to starch content, with foods containing a high sugar to starch content to reach a target ratio of starch to sugar 1: 1.2.
- Low Sugar Diet (12 Weeks) in Controls: A low sugar (10% total energy), high starch diet was provided by the exchange of 66% of the participants daily intake of carbohydrate. This was achieved by replacing foods with a high sugar to starch content, with foods containing a low sugar to starch content to reach a target ratio of starch to sugar of 5:1.
Arm/Group | High Sugar Diet (12 Weeks) in Men With NAFLD | Low Sugar Diet (12 Weeks) in Men With NAFLD | High Sugar Diet (12 Weeks) in Controls | Low Sugar Diet (12 Weeks) in Controls
Number analyzed (Participants) | 11 | 11 | 14 | 14
grams/day | 20.9 (2.1) | 18.9 (2.1) | 16.6 (1.4) | 12.4 (1.2)
Statistical Analysis 1: Comparison: High Sugar Diet (12 Weeks) in Men With NAFLD vs Low Sugar Diet (12 Weeks) in Men With NAFLD vs High Sugar Diet (12 Weeks) in Controls vs Low Sugar Diet (12 Weeks) in Controls; The sample size of the NAFDL & Control groups was based on primary outcome measures for a trace-labelling study of VLDL kinetics (VLDL1 apo B & TAG production rates). From the literature there was an 80% probability that our study will detect a difference in the production rates of VLDL1 apo B of 30% (α=39%), and 26% for VLDL1-TAG (α=33%). A paired comparison of two diets (5% level), gave sample sizes of n=15 for each group. Note: All reported P-values were calculated; Test type: Other; p < 0.05, Mixed Models Analysis — Outcome measures were analysed as dependent variables in a general linear mixed model. All outcome variables in the model analysed were part of an priori hypothesis, and for this reason were not subject to adjustment for multiple comparisons; Mixed model analysis was appropriate for testing differences between 2 Groups on 2 Diets (NAFLD, Control,high & low sugar diets); General linear mixed model = 2 — Details of our statistical approach are given below; For outcome measures for which there were four samples from each participant (pre- and post-diets, for each period), the post-diet measurements were analysed as dependent variables in a general linear mixed model, with the following fixed categorical, non-random, explanatory effects: period, treatment (low and high sugar diet), period by treatment interaction (to detect carry-over effects), liver fat level (NAFLD and Control) and treatment by liver fat level interaction. The pre-diet measurements for each period, and bodyweights (pre- and post-diets) were included as covariates in the model, with participant as a model random effect. For outcome measures for which there were two samples for each participant (post-diets; end of each dietary intervention period only), each measurement for the combined groups (NAFLD and controls), for the 2-period cross-over, were analysed in a general linear mixed model with the same fixed categorical effects and bodyweights as covariates

2. Primary Outcome: Production Rate VLDL-1 Apoprotein B
Description: The in vivo production rate of VLDL-1 apoprotein B, trace-labelled with [I-13C] leucine (leucine with carbon-13), measured in units of milligrams/day.
Time Frame: After (post-diet) two 12 week diets (high sugar versus low sugar) in men with NAFLD (n=11) versus Controls (n=14)
Population: Population consisted of two groups: Group 1: NAFLD; men with raised liver fat ( >5%), n=11. Group 2: Controls; men with low liver fat (<5%) n=14.
Measure: Mean (Standard Error); unit: mg/day
Groups:
- Low Sugar Diet (12 Weeks) in Men With NAFLD: A low sugar (9% total energy), high starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with a high sugar to starch content, with foods containing a low sugar to starch content to reach a target ratio of starch to sugar of 5:1
- Low Sugar Diet (12 Weeks) in Controls: A low sugar (10% total energy), high starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with a high sugar to starch content, with foods containing a low sugar to starch content to reach a target ratio of starch to sugar of 5:1
Arm/Group | High Sugar Diet (12 Weeks) in Men With NAFLD | Low Sugar Diet (12 Weeks) in Men With NAFLD | High Sugar Diet (12 Weeks) in Controls | Low Sugar Diet (12 Weeks) in Controls
Number analyzed (Participants) | 11 | 11 | 14 | 14
mg/day | 481 (76) | 492 (58) | 546 (56) | 414 (54)
Statistical Analysis 1: Comparison: High Sugar Diet (12 Weeks) in Men With NAFLD vs Low Sugar Diet (12 Weeks) in Men With NAFLD vs High Sugar Diet (12 Weeks) in Controls vs Low Sugar Diet (12 Weeks) in Controls; The sample size for NAFLD & Control groups was based on primary outcome measures for a trace-labelling study of VLDL kinetics (VLDL1 apo B and triacylglycerol production rates). From the literature there was an 80% probability that our study will detect a difference in the production rates of VLDL1 apo B of 30% (α=39%), and 26% for VLDL1-TG (α=33%). A paired comparison of two diets (5% level) produced sample sizes of n=15 for each group. Note: All reported P-values were calculated; Test type: Other; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mixed model analysis was appropriate for testing the impact of 'Diet' (high and low sugar) and Group (NAFLD and Control) status on outcome variables; General linear mixed model = 11 — Details of our statistical analyses are given below; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Kinetics of Systemic Non-esterified Fatty Acids by [C-13]-Trace-labelled Palmitate
Description: Palmitate was labelled in vivo by the infusion of [U-13 carbon]. This provides a measure of the rate of intra-cellular lipolysis and contribution of systemic palmitate to the synthesis of triacylglycerol in the liver in units of micro mols/L (umol/L).
Time Frame: After (post-diet) two 12 week diets (high sugar versus low sugar) in men with NAFLD (n=11) versus Controls (n=14)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: umol/L
Groups:
- High Sugar Diet (12 Weeks) in Men With NAFLD: A high sugar diet (27% total energy), low starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with low sugar to starch content, with foods containing a high sugar to starch content to reach a target ratio of starch to sugar of 1:1.2
- High Sugar Diet (12 Weeks) in Controls: A high sugar diet (28% total energy), low starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with low sugar to starch content, with foods containing a high sugar to starch content to reach a target ratio of starch to sugar of 1:1.2.
- Low Sugar Diet (12 Weeks) in Controls: A low sugar (9% total energy), high starch diet was provided by the exchange of 66% of the participants daily intake of carbohydrate. This was achieved by replacing foods with a high sugar to starch content, with foods containing a low sugar to starch content to reach a target ratio of starch to sugar of 5:1.
Arm/Group | High Sugar Diet (12 Weeks) in Men With NAFLD | Low Sugar Diet (12 Weeks) in Men With NAFLD | High Sugar Diet (12 Weeks) in Controls | Low Sugar Diet (12 Weeks) in Controls
Number analyzed (Participants) | 11 | 11 | 14 | 14
umol/L | 169 (11) | 147 (12) | 168 (15) | 168 (17)
Statistical Analysis 1: Comparison: High Sugar Diet (12 Weeks) in Men With NAFLD vs Low Sugar Diet (12 Weeks) in Men With NAFLD vs High Sugar Diet (12 Weeks) in Controls vs Low Sugar Diet (12 Weeks) in Controls; The sample size of the NAFDL & Control groups was based on primary outcome measures for a trace-labelling study of VLDL kinetics (VLDL1 apo B & TAG production rates). From the literature there was an 80% probability that our study will detect a difference in the production rates of VLDL1 apo B of 30% (α=39%), and 26% for VLDL1-TG (α=33%). A paired comparison of two diets (5% level), gave sample sizes of n=15 for each group. Note: All reported P-values were calculated; Test type: Other; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; General linear mixed model = 110 — Details of our statistical analyses are given below; [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: De Novo Lipogenesis (Rate of Triacylglycerol (TAG) Synthesis in the Liver) as Measured by Contribution to VLDL-1 TAG Production Rate
Description: Acetyl CoA (Co-enzyme-A) is labelled in vivo by the consumption of [2H20] (2H20=deuterated 'heavy'-labelled water). Recovery and detection of this label in VLDL-1 by GC-MS (Gas Chromatography-Mass Spectrometry), provides a measure of fatty acid and TAG synthesis in the liver in terms of its contribution to the production rate of VLDL-1 TAG in units of grams/day.
Time Frame: After (post-diet) two 12 week diets (high sugar versus low sugar) in men with NAFLD (n=11) versus Controls (n=14)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: grams/day
Groups:
- High Sugar Diet (12 Weeks) in Men With NAFLD: A high sugar (27%), low starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with low sugar to starch content, with foods containing a high sugar to starch content to reach a target ratio of starch to sugar of 1:1.2
- Low Sugar Diet (12 Weeks) in Men With NAFLD: A low sugar (9%), low starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with a high sugar to starch content, with foods containing a low sugar to starch content to reach a target ratio of starch to sugar of 5:1
- High Sugar Diet (12 Weeks) in Controls: A high sugar (28%), low starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with low sugar to starch content, with foods containing a high sugar to starch content to reach a target ratio of starch to sugar of 1:1.2
- Low Sugar Diet (12 Weeks) in Controls: A low sugar (10%), low starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with a high sugar to starch content, with foods containing a low sugar to starch content to reach a target ratio of starch to sugar of 5:1
Arm/Group | High Sugar Diet (12 Weeks) in Men With NAFLD | Low Sugar Diet (12 Weeks) in Men With NAFLD | High Sugar Diet (12 Weeks) in Controls | Low Sugar Diet (12 Weeks) in Controls
Number analyzed (Participants) | 11 | 11 | 14 | 14
grams/day | 1.66 (0.39) | 1.59 (0.34) | 1.32 (0.43) | 0.56 (0.14)
Statistical Analysis 1: Comparison: High Sugar Diet (12 Weeks) in Men With NAFLD vs Low Sugar Diet (12 Weeks) in Men With NAFLD vs High Sugar Diet (12 Weeks) in Controls vs Low Sugar Diet (12 Weeks) in Controls; [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; General linear mixed model = 0.26 — Details of our statistical approach are given below; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: Intra-hepatocellular Lipid (IHCL) or % Liver Fat
Description: Percentage of intra-hepatocellular lipid (IHCL or % liver fat) was measured by magnetic resonance spectroscopy (MRS).
Time Frame: After (post-diet) two 12 week diets (high sugar versus low sugar) in men with NAFLD (n=11) versus Controls (n=14)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percentage of liver fat
Groups:
- High Sugar Diet (12 Weeks) in Men With NAFLD: A high sugar (27% total energy), low starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with low sugar to starch content, with foods containing a high sugar to starch content to reach a target ratio of starch to sugar of 1:1.2.
- High Sugar Diet (12 Weeks) in Controls: A high sugar (28% total energy), low starch diet was provided by the exchange of two thirds of the participants daily intake of carbohydrate. This was achieved by exchanging foods with low sugar to starch content, with foods containing a high sugar to starch content to reach a target ratio of starch to sugar of 1:1.2.
Arm/Group | High Sugar Diet (12 Weeks) in Men With NAFLD | Low Sugar Diet (12 Weeks) in Men With NAFLD | High Sugar Diet (12 Weeks) in Controls | Low Sugar Diet (12 Weeks) in Controls
Number analyzed (Participants) | 11 | 11 | 14 | 14
Percentage of liver fat | 24.2 (6.8) | 14.2 (3.2) | 3.6 (1.3) | 1.5 (0.3)
Statistical Analysis 1: Comparison: High Sugar Diet (12 Weeks) in Men With NAFLD vs Low Sugar Diet (12 Weeks) in Men With NAFLD vs High Sugar Diet (12 Weeks) in Controls vs Low Sugar Diet (12 Weeks) in Controls; [analysis description as in outcome 3, analysis 1]; Test type: Other; p > 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; General linear mixed model = 10 — Details of our statistical analyses are described below; [other analysis details as in outcome 1, analysis 1]

6. Secondary Outcome: Plasma Concentration of Triacylglycerol
Description: Plasma concentration of triacylglycerol (TAG) was measured in the post-absorptive state (after 12h fast) and expressed in units of mmol/L (shown as log transformed geometric means)
Time Frame: After (post-diet) two 12 week diets (high sugar versus low sugar) in men with NAFLD (n=11) versus Controls (n=14)
Population: as for outcome 2
Measure: Geometric Mean (Standard Error); unit: mmol/L
Arm/Group | High Sugar Diet (12 Weeks) in Men With NAFLD | Low Sugar Diet (12 Weeks) in Men With NAFLD | High Sugar Diet (12 Weeks) in Controls | Low Sugar Diet (12 Weeks) in Controls
Number analyzed (Participants) | 11 | 11 | 14 | 14
mmol/L | 2.05 (0.24) | 1.77 (0.22) | 1.33 (0.15) | 1.13 (0.08)
Statistical Analysis 1: Comparison: High Sugar Diet (12 Weeks) in Men With NAFLD vs Low Sugar Diet (12 Weeks) in Men With NAFLD vs High Sugar Diet (12 Weeks) in Controls vs Low Sugar Diet (12 Weeks) in Controls; [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; General linear mixed model = 0.28 — Details of our statistical analyses are given below; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- High Sugar Diet in NAFLD Men (n=11): A high sugar (27% total energy), low starch diet was provided by the exchange of 66% of the participants daily intake of carbohydrate. This was achieved by exchanging foods with a low sugar to starch content, with foods containing a high sugar to starch content to reach a target ratio of starch to sugar 1: 1.2.
- Low Sugar Diet in NAFLD Men (n=11): A low sugar (9% total energy), high starch diet was provided by the exchange of 66% of the participants daily intake of carbohydrate. This was achieved by replacing foods with a high sugar to starch content, with foods containing a low sugar to starch content to reach a target ratio of starch to sugar of 5:1.
- High Sugar Diet in Controls (n=14): A high sugar (28% total energy), low starch diet was provided by the exchange of 66% of the participants daily intake of carbohydrate. This was achieved by exchanging foods with a low sugar to starch content, with foods containing a high sugar to starch content to reach a target ratio of starch to sugar 1: 1.2.
- Low Sugar Diet in Controls (n=14): A low sugar (10% total energy), high starch diet was provided by the exchange of 66% of the participants daily intake of carbohydrate. This was achieved by replacing foods with a high sugar to starch content, with foods containing a low sugar to starch content to reach a target ratio of starch to sugar of 5:1.
Arm/Group | High Sugar Diet in NAFLD Men (n=11) | Low Sugar Diet in NAFLD Men (n=11) | High Sugar Diet in Controls (n=14) | Low Sugar Diet in Controls (n=14)
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
A limitation of metabolic studies is their small sample size, which is a consequence of the invasive nature, extent, labour intensity, and high cost ($850,000) of the metabolic investigations e.g. infusion/ingestion of 4 stable isotope tracers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes